CLINICAL TRIAL: NCT05627466
Title: Expanded Access Program for Magrolimab
Brief Title: US Expanded Access Program for Magrolimab in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: No longer available | Type: Expanded Access
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-546-6531
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — magrolimab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously
  Other Names: GS-4721

SUMMARY:
The goal of this expanded access program is to provide rapid access to magrolimab free-of-cost material, to treat patients in the United States suffering from relapsed or refractory acute myeloid leukemia (AML).

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals with confirmation of acute myeloid leukemia (AML) according to WHO 2016 classification who are refractory or relapsed, ineligible for all known drugs with proven efficacy, and ineligible for existing clinical studies; and the treating physician has assessed that the potential benefits of magrolimab outweigh the risks.
* Eastern Cooperative Oncology Group performance status score of 0 to 3.
* Treating physician plans to administer magrolimab in combination with azacitadine/venetoclax or magrolimab in combination with azacitadine alone, following the indication-specific combinations described in the protocol.

Key Exclusion Criteria:

* Known hypersensitivity to magrolimab, azacitidine, venetoclax, their metabolites, or formulation excipients, if applicable to planned treatment regimen.
* Prior treatment with cluster of differentiation (CD)47 or signal regulatory protein alpha (SIRPα)-targeting agents.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences

REFERENCES:
- See also: Click on this link to request access through the Bionical Emas Patient Access Portal — http://www.yourpatientaccess.com
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-546-6531